CLINICAL TRIAL: NCT04833387
Title: PD-1 Antibody as a Sequential Therapy Following Preoperative Chemoradiotherapy for Locally Advanced pMMR/MSS Rectal Cancer: an Open, Multi-center, Phase II Clinical Trial
Brief Title: PD-1 Antibody Following Preoperative Chemoradiotherapy for Locally Advanced pMMR/MSS Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-092
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: PD-1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 antibody + capecitabine + radiation (Experimental)
  Interventions: Drug: PD-1 antibody

INTERVENTIONS:
Drug: PD-1 antibody — Capecitabine:Dose of 1650mg/m2,14days; Radiation:50Gy/25 fractions;IBI308: 200mg on day1 of each cycle, 3 cycles; Surgical therapy:The resection (LAR), intersphincteric resection (ISR), or abdominoperineal resection (APR)

SUMMARY:
In this open-label phase II study, patients will be scheduled for neoadjuvant treatment with PD-1 antibody following preoperative Chemoradiotherapy with capecitabine for pMMR/MSS rectal cancer staged as locally advanced (cT3-T4N+/-M0 for rectal cancer). This treatment will be given during the window period until surgical resection of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients who personally provided written consent for participation in the study
* Treatment-naive patients with rectal cancer, in whom the inferior margin of the tumor was at a distance of 12 cm or less from the AV before CRT
* Primary rectal cancer histopathologically confirmed to be adenocarcinoma
* Clinical stage of T3,and T4 ,N any,M0,before CRT
* Macroscopic radical resection could be feasible, based on diagnostic imaging before CRT
* Patients with the ECOG performance status of 0 or 1 at the time of enrollment
* Patients without distant metastasis on the imaging test before CRT
* Preoperative biopsy of tumor immunohistochemistry TPS>1% or CPS>1
* Life expectancy of greater than 2 years
* No signs of intestinal obstruction; or the obstruction has been relieved after the proximal colostomy operation
* Hematology: WBC>4000/mm3; PLT>100000/mm3; Hb>10g/dL
* Liver function: SGOT and SGPT are less than 1.5 times the normal value; bilirubin is less than 1.5mg/dL
* Renal function: creatinine <1.8mg/dL Others: non-pregnant or breast-feeding women; no other malignant diseases (except for non-melanoma or cervical carcinoma in situ) within 5 years or during the same period; no mental illness that causes the inability to obtain informed consent; no other serious diseases that can shorten the survival time disease.
* Have not received rectal surgery in the past;
* Have not received chemotherapy or radiotherapy in the past;
* Have not received biological treatment in the past;
* Past endocrine therapy: unlimited.

Exclusion Criteria:

* Rectal cancer with unstable microsatellite (MSI or dMMR);
* Preoperative biopsy of tumor immunohistochemistry TPS≤1% or CPS≤1
* Known history of human immunodeficiency virus (HIV) or chronic hepatitis B or C (high copy viral DNA);
* Autoimmune diseases;
* Other active clinical serious infections (>NCI-CTC version 3.0);
* Patients in clinical phase I;
* There is evidence that there is distant metastasis before surgery;
* Cachexia, decompensation of organ function;
* Have a history of pelvic or abdominal radiotherapy;
* Multiple primary cancers;
* Patients who need treatment for seizures (such as steroids or anti-epileptic treatment);
* Have a known additional malignant tumors within 5 years. Exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
* Chronic inflammatory bowel disease, intestinal obstruction;
* Drug abuse and medical, psychological or social conditions may interfere with patients' participation in research or have an impact on the evaluation of research results;
* Known or suspected to be allergic to the study drug or to any drug given in connection with this test;
* Any unstable conditions or situations that may endanger patient safety and compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 1 year
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | 3 years
Overall survival (OS) | 3 years
Clinical complete response (CCR) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou Z, Liao L, Xiao W, Sui Q, Han K, Xiao B, Li Y, Mei W, Yu J, Hong Z, Chen Q, Song R, Li D, Zhang X, Wang Q, Pan Z, Jiang W, Ding P. Neoadjuvant chemoradiotherapy plus sintilimab in pMMR/MSS rectal cancer patients with PD-L1 TPS >/= 1% or CPS >/= 1: an open-label, prospective, phase II study. NPJ Precis Oncol. 2025 Jul 12;9(1):237. doi: 10.1038/s41698-025-01018-0. PMID 40652024